CLINICAL TRIAL: NCT05097950
Title: Labor Induction and Pain Relief Prior to Insertion of a Balloon Catheter
Brief Title: Labor Induction and Pain Relief With Paracetamol Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Inshirah Sgayer, inshirah sgayer, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0065-21-NHR
Record Dates: First submitted 2021-09-12; First posted 2021-10-28 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Administration of 1 gr paracetamol I.V
  Interventions: Drug: Administration of 1 gr paracetamol I.V
- Control Group (Placebo Comparator): Administration of 100 ml. sodium chloride 0.9% IV
  Interventions: Drug: Administration of 1 gr paracetamol I.V

INTERVENTIONS:
Drug: Administration of 1 gr paracetamol I.V — Administration of 1 gr paracetamol I.V

SUMMARY:
Single-blind study conducted on 2 randomly selected groups of pregnant women carrying a single fetus (from week 37 onward). One group will receive paracetamol 1 gr I.V. prior to insertion of balloon catheter and the control group will receive 100 ml sodium chloride 0.9% I.V prior to insertion of balloon catheter. An assessment of pain management will be conducted using various assessment tools. additionally, mode of delivery and time from catheter insertion to delivery will be assessed.

DETAILED DESCRIPTION:
Single-blind study conducted on 2 randomly selected groups of pregnant women carrying a single fetus (from week 37 onward). One group will receive paracetamol 1 gr I.V. prior to insertion of balloon catheter and the control group will receive 100 ml sodium chloride 0.9% I.V prior to insertion of balloon catheter.

assessment of pain during catheter balloon insertion will be assessed using visual analogue scale (VAS) instrument with scores 1 to 10.

An assessment of pain management will also be conducted using various assessment tools:

1. Brief Pain Inventory short form (BPIsf) - before balloon insertion and at various time intervals.
2. Hospital Anxiety and Depression Scale (HADS) - 1 hr. before balloon insertion and immediately upon removal of catheter.
3. Patient Experience Questionnaire - upon transfer to delivery room.
4. Socio-demographic Questionnaire

Additionally, obstetrics outcomes will be recorded including time from catheter to delivery, mode of delivery. these parameters will be compared between the two groups (those who recieved paracetamol versus normal saline 0.9%).

ELIGIBILITY:
Inclusion Criteria:

Women from 18-44 yrs of age 37 weeks pregnant and onward singleton pregnancy induction of labor using a balloon catheter Nulliparity

Exclusion Criteria:

1. Sensitivity to paracetamol.
2. Past Cesarean section
3. Multiple pregnancy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 141 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
PAIN assessment during catheter balloon insertion | through study completion, an average of 1 year
  pain assessment during catheter balloon insertion will be conducted using Visual Analogue Scale (VAS) instruments with scores from 10 to 10
maternal satisfaction | through study completion, an average of 1 year
  maternal satisfaction will be evaluated using a questionnaire

SECONDARY OUTCOMES:
need for additional analgesic agent | through study completion, an average of 1 year
  need for additional analgesic agent than paracetamol after catheter balloon insertion
maternal mobility | through study completion, an average of 1 year
  women were asked through a questionnaire about whether they were immoblile after the catheter insetion using a score from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Inshirah Sgayer, Nahariya, Israel